CLINICAL TRIAL: NCT02399462
Title: Acthar for Treatment of Post-transplant FSGS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding terminated prematurely
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0999; ACTH-101 (Other: UNC)
Record Dates: First submitted 2015-01-08; First posted 2015-03-26 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: FSGS; Renal Transplantation; Kidney Transplantation
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Drug Arm (Experimental): Acthar SC injections
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — Agent Dose Route Schedule H.P. Acthar Gel 40 units SC twice weekly* Weeks 1 and 2
  H.P. Acthar Gel 80 units SC twice weekly* Weeks 3 through 24
  H.P. Acthar Gel 80 units SC once weekly* Weeks 25 through 26
  H.P. Acthar Gel 40 units SC once weekly* Weeks 27 through 28
  *Injections are to be spaced 72-96 hours apart (+/-6 hours).
  Other Names: ACTH (adrenocorticotropic hormone ), corticotropin

SUMMARY:
This is an open label safety and feasibility trial using Acthar® in addition to center-specific standard therapy including plasma exchange, for treatment of post transplant recurrent FSGS and post transplant recurrent idiopathic membranous nephropathy. Subjects will receive Acthar® 40 units subcutaneously (SC) twice weekly for two weeks then 80 units SC twice weekly for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Proteinuria > 1 g/d by urine protein/creatinine ratio (UP/C) or 24 hour urine collection
* If treated with an angiotensin-converting-enzyme inhibitor (ACEi) or Angiotensin II receptor blockers (ARB), must be on a stable dose for at least 2 weeks prior to enrollment
* Newly diagnosed recurrent focal and segmental glomerulosclerosis (FSGS), or current/previous treatment of recurrent FSGS with no evidence of at least a partial response as defined by one or more of the following:

  1. Recurrent FSGS confirmed by renal transplant biopsy (FSGS on light microscopy and/or foot process effacement on electron microscopy), with FSGS as the primary disease confirmed by native renal biopsy prior to transplant
  2. FSGS confirmed by renal transplant biopsy (FSGS on light microscopy and/or foot process effacement on electron microscopy), within 18 months post transplant
  3. Patients at any time period post transplant with an established diagnosis of recurrent FSGS in the first 18 months post transplant who did not respond to conventional therapy as defined by persistent proteinuria of > 3 g/d by UP/C or 24 hour urine collection

Exclusion Criteria:

* Lactation, pregnancy or refusal of birth control in women of childbearing potential
* Infection with human immunodeficiency virus (HIV), hepatitis B, hepatitis C, or parvovirus B-19
* Malignancy (with the exception of treated and cured basal cell or squamous cell carcinoma)
* Evidence of diabetic nephropathy, transplant glomerulopathy or other pathologies that could be associated with secondary FSGS on renal transplant biopsy
* Non-renal organ transplant (with the exception of pancreas transplant)
* Contraindication to receiving Acthar®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
number of patients with proteinuria | 24 and 52 weeks
  partial and complete remission of proteinuria

SECONDARY OUTCOMES:
Graft loss | during study period
  graft loss defined by return to dialysis, re-transplant or death during study period
eGFR change | weeks 4,8,12,16,20 and 24
  estimated Glomerular filtration rate (eGFR MDRD formula) change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Karin True, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No